CLINICAL TRIAL: NCT04396444
Title: Lavender Aromasticks as an Option for Pain Control in the Vascular Surgery Population
Brief Title: Lavender Aromasticks for Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: dōTERRA International (Industry)
Responsible Party: Principal Investigator, Rebecca Hornberger, Clinical Nurse, Heart and Vascular Progressive Care Unit, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00011852
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Pain Perception; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Aromastick Group (Experimental): The aromastick is a plastic tube, similar in size to a lipstick. A study team member will prepare the aromastick by infusing ten drops of lavender essential oil onto a blank cotton wick inside the tube and sealing the cap.
  Interventions: Combination Product: Aromastick
- Blank Aromastick Group (Placebo Comparator): A study team member will prepare the blank aromastick by placing a blank cotton wick inside the aromastick tube and sealing the cap.
  Interventions: Combination Product: Aromastick

INTERVENTIONS:
Combination Product: Aromastick — Vascular surgery patients will be randomized to either the intervention group and receive a lavender infused aromastick to use as an adjunct to their inpatient pain management plan, or to the control group, given a blank aromastick. Subjects will be blinded to their group.

SUMMARY:
The purpose of this randomized pilot study is to collect preliminary data on the impacts of lavender essential oil aromatherapy on the patient-reported quality of pain management provided for the vascular surgery patient population. The investigators hypothesize that individuals who use a lavender aromastick as a part of their pain management plan will report improved perceptions of the quality of their pain management as measured by the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R).

Subjects will be randomized to the control (empty aromastick) and intervention group (aromastick infused with lavender oil), and will use this device as an addition to their pain management plan.

Additionally, this pilot study will allow the researchers to evaluate the feasibility of a larger randomized control trial, assess the validity of the survey tool, and collect feedback from patients on the acceptability of the aromatherapy intervention as a complementary therapy during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 and over admitted to the vascular surgery service line on the Heart and Vascular Progressive Care Unit (HVPCU)
2. Not cognitively impaired
3. Able to perform teach-back of the education regarding safe use of the aromastick
4. Able to demonstrate use of the Numeric Pain Rating Scale (NPRS), as evidenced by their ability to answer the initial NPRS question on the Adult Admission II Form used to admit all patients to the hospital
5. English is the primary language, as identified by the Adult Admission II Form

Exclusion Criteria:

1. Subjects who are unable to consent themselves
2. Subjects who cannot provide teach-back on the safe use of the aromastick
3. Subjects unable to use the NPRS to rate their pain
4. Research team member and/or bedside nurse assess that subject has a cognitive deficit that would prohibit safe use of the aromastick
5. Subjects on suicide precautions
6. Pregnant subjects
7. Prisoners
8. Individuals under age 18
9. Subjects with a current plan to use personal aromatherapy devices during their inpatient stay
10. Subjects with known lavender allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoints for this study are patients' self-reported evaluations of the quality of pain management provided during their hospital stay. | Measured on day 6 of hospital stay or day of discharge; whichever is sooner
  Measured using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) survey tool. The APS-POQ-R has 18 primary questions with continuous rating scales from 0 - 10 or from 0% - 100%. This study, with permission from the original authors, uses a modified survey, with 10 questions evaluating the subject's pain levels and degree to which pain interferes with various aspects of their quality of life. In these questions, higher numbers indicate higher levels of pain and distress. Four additional Likert style questions evaluate subjects' satisfaction with pain management, with higher numbers indicating higher levels of satisfaction.

SECONDARY OUTCOMES:
Subjects' evaluation of the aromastick | Measured on day 6 of hospital stay or day of discharge; whichever is sooner
  Survey questions will also be asked about use of the aromastick to evaluate acceptability of the intervention device. These are yes/no questions, and questions measuring the frequency of device use.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hornberger, MSN, Principal Investigator — Penn State Health Milton S Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon DB, Polomano RC, Pellino TA, Turk DC, McCracken LM, Sherwood G, Paice JA, Wallace MS, Strassels SA, Farrar JT. Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) for quality improvement of pain management in hospitalized adults: preliminary psychometric evaluation. J Pain. 2010 Nov;11(11):1172-86. doi: 10.1016/j.jpain.2010.02.012. Epub 2010 Apr 18. PMID 20400379